CLINICAL TRIAL: NCT03933423
Title: Using Community Health Workers and In-home LED Phototherapy to Dramatically Reduce Brain Damage From Neonatal Jaundice in Low to Middle Income Countries: A Feasibility Trial
Brief Title: Home Based Phototherapy for Neonatal Jaundice
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: International Centre for Diarrhoeal Disease Research, Bangladesh (Other)
Collaborators: Stanford University (Other); Dhaka Shishu Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PR-19004
Record Dates: First submitted 2019-04-23; First posted 2019-05-01 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Neonatal Jaundice
MeSH Terms: conditions — Jaundice, Neonatal | interventions — Mass Screening

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Active Comparator): Educational session of pregnant mothers, blood grouping of parents and identifying risk factors for developing jaundice, screening newborns for neonatal jaundice, glucose 6-phosphate dehydrogenase deficiency and illness, Home based phototherapy and referral.
  Interventions: Device: Home based phototherapy and referral
- Control (No Intervention): No intervention will be deliver

INTERVENTIONS:
Device: Home based phototherapy and referral — CHWs will visit the household twice in a month and will counsel mother and families on use of preventive care such as routine antenatal check care and newborn care. The investigators will conduct blood grouping and rhesus (Rh) typing. If the mother is Rh negative, investigators will also measure the Rh status of the father prior to delivery to determine the risk of Rh disease in the newborn. The investigators will establish an emergency contact system both in intervention and comparison arm where mothers and family members contact and inform the research team about delivery. The trained phlebotomist will collect cord blood for measuring glucose 6-phosphate dehydrogenase and infant blood type, Rh status, direct antigen testing. The investigators will develop a protocol for treating infants at home based on the ETAT (Emergency Triage Assessment AND Treatment) AAP (American Academy of Paediatrics) guidelines and treat with LED based phototherapy
  Other Names: Educational session, identifying risk factors and, screening
  Arms: Intervention

SUMMARY:
The main purpose of the study is to deliver community health worker based prevention, early screening and management of neonatal Jaundice using battery powered LED phototherapy device at the household level.

DETAILED DESCRIPTION:
Bangladesh like other low and middle-income countries has a high burden of hyperbilirubinemia induced neonatal morbidity and mortality. Approximately 60%-80% of newborns develop neonatal jaundice and 18% of infants are at risk for adverse outcomes from neonatal jaundice. Severe neonatal jaundice can put neonates at risk for long term neuro-developmental impairments and death. Delay in diagnosis and treatment of severe neonatal jaundice can result in brain damage to the newborn that is preventable with timely treatment.

Approximately 14 million infants per year in low to middle-income countries (LMIC) are at risk from neonatal jaundice progressing to extreme hyperbilirubinemia and brain damage. Nearly 80% of the 481,000 cases of extreme hyperbilirubinemia are in LMIC because infants are identified too late or health facility treatment is inaccessible or inadequate.

New, low-cost, easy to use screening and phototherapy treatment technologies enable our proposed redesign of care delivery in LMIC to save infant's brains. The investigators plan to shift care from specialists and hospitals to community health workers (CHW) and homes. Investigators will integrate CHW-led prevention during pregnancy, with timely household screening and treatment. Investigators will reach infants before brain damage occurs and treat infants who would not otherwise be treated.

LMIC including Bangladesh have had difficulty addressing neonatal jaundice because of the expense and logistics of providing timely prevention, screening and treatment to families. This study aim to test 3 hypothesis:

H1: Prenatal modules for pregnant mothers will increase breastfeeding rates at 1 hour of life and at 3 months of age.

H2: CHWs can screen 80% of newborns by 48 hours of age for jaundice and are skilled in identifying sick infants.

H3: CHW-led household screening for neonatal jaundice will increase the rate of indicated treatment for neonatal jaundice compared to current practice.

Investigators will conduct formative research to engage Government and other stakeholders to develop intervention package for prevention and treatment of neonatal jaundice and configuring and adapting LED phototherapy device to use for home treatment. Investigators will then conduct randomized control trial to implement the intervention package in intervention community and will assess the effectiveness of the intervention package. Investigators will compare the rates of indicated treatment for neonatal jaundice in the intervention and treatment arms.

ELIGIBILITY:
Inclusion Criteria:

* The mothers are at late 2nd or early 3rd trimester of their pregnancy and agreed to enroll as study participants
* They are planning to stay in the study village for the next 12 months (if a mother is planning to give birth at her natal home and then return, she will still not be a candidate for enrollment)

Exclusion Criteria:

* Pregnant mother with confirmed multiple pregnancy.
* Pregnant mother with medically identified psychological disorder.
* Any known maternal danger sign.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Pregnant mothers above 18 years
Enrollment: 500 (Estimated)
Dates: Start 2019-05-01 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Breastfeeding rates within 1 hour of age | 6-8 months after the intervention
  Mother reported breastfeeding rates within 1 hour of age will be measured following structured survey
Breastfeeding rates upto 3 months of age | 6-8 months after the intervention
  Mother reported breastfeeding rates after 3 months of age will be measured following structured survey
Number of newborns having at least one postnatal check-up within 48 hours. | 6-8 months after the intervention
  This measurement will be taken within 2 months of child birth through a structured survey, reported by mother.
Number of newborns screened for neonatal jaundice | 6-8 months after the intervention
  Number of newborns screened for neonatal jaundice either in home or any government or non-government health facilities within 7 days of birth through a structured survey reported by mother.
Number of newborns that received indicated treatment for neonatal jaundice | 6-8 months after the intervention
  Number of children receiving indicated treatment for neonatal jaundice either in home or health facilities will be measured by a mother reported structured survey after 2 months of child birth
Community health workers (CHW's) skill in assessing sick newborns | During 6-8 months of the intervention
  CHW's skill will be measured through a structured observation following a check list and subjective and objective assessment by registered physician

CONTACTS AND LOCATIONS:
Locations (1):
- Mirzapur, Tāngāil, Dhaka Division, Bangladesh

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Jahan F, Foote E, Rahman M, Shoab AK, Parvez SM, Nasim MI, Hasan R, El Arifeen S, Billah SM, Sarker S, Hoque MM, Shahidullah M, Islam MS, Ashrafee S, Darmstadt GL. Evaluation of community health worker's performance at home-based newborn assessment supported by mHealth in rural Bangladesh. BMC Pediatr. 2022 Apr 22;22(1):218. doi: 10.1186/s12887-022-03282-6. PMID 35459113